CLINICAL TRIAL: NCT05866562
Title: Dupilumab in the Treatment of Pediatric Alopecia Areata
Acronym: PEDAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Emma Guttman, Waldman Professor and System Chair, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-00744
Record Dates: First submitted 2023-02-22; First posted 2023-05-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Experimental): 200 mg or 300 mg SC injections every 2 or 4 weeks (weight based)
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Injections without active ingredients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Participants weighing 15 kg < 30 kg = 300 mg Every 4 Weeks; Participants weighing 30 kg < 60 kg = 200 mg Every 2 Weeks; Participants weighing ≥ 60 kg = 300 mg Every 2 Weeks;
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Placebo — Participants weighing 15 kg < 30 kg Every 4 Weeks; Participants weighing 30 kg < 60 kg Every 2 Weeks; Participants weighing ≥ 60 kg Every 2 Weeks
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled clinical trial. The study will take place at four sites. This trial will enroll a total of 76 children and adolescents with moderate to severe AA (affecting at least 30% of the scalp) at the time of screening with a targeted 61 participants completing through Week 48. All subjects must have evidence of hair regrowth within the last 7 years of their last episode of hair loss; and have screening IgE ≥200 and/or have personal and/or familial history of atopy.

Study participation will be up to 124 weeks, consisting of: a screening period of up to 4 weeks; a 48-week placebo-controlled period; a 48-week open-label extension period; followed by a 24-week follow-up period.

DETAILED DESCRIPTION:
After providing consent, subjects will be assessed for study eligibility during the screening period (within 4 weeks of Baseline), which includes a review of past and current medical conditions, detailed review of past and current medications, a physical examination, clinical assessments, and laboratory tests for safety. Subjects who meet inclusion and exclusion criteria for eligibility will undergo Baseline assessments at Week 0. Subjects will return for visits every 8-16 weeks for repeat clinical assessments, medication reviews, and monitoring for adverse events. Female subjects will undergo a urine pregnancy test (where applicable) at each of these visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who are at least 6 years old and under 18 years old, who can provide assent (if appropriate), and for whom signed informed consent can be provided by parent or legal guardian prior to participation in any study assessments or procedures

  -- Participant is able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product (IP), FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

  * Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR
  * Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]);
* Participant has a history of at least 6 months of moderate to severe AA (≥ 50% scalp involvement) as measured using the SALT score.
* Participant has a screening IgE ≥ 200 and/or personal and/or familial history of atopy (including asthma, atopic dermatitis, allergic rhinitis, food allergy, or eosinophilic esophagitis)
* Participant is judged to be in otherwise good overall health following a detailed medical and medication history, physical examination, and laboratory testing.

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Participant is pregnant or breastfeeding.
* Participant's cause of hair loss is indeterminable and/or they have concomitant causes of alopecia, such traction, cicatricial, pregnancy-related, drug-induced, telogen effluvium, or advanced androgenetic alopecia (i.e. Ludwig Type III or Norwood-Hamilton Stage ≥ V).
* Participant has a history of AA with no evidence of hair regrowth for ≥ 7 years since their last episode of hair loss.
* Severe, uncontrolled asthma (having 2 or exacerbations in the last 12 months that require systemic steroids and/or hospitalization) or a history of life-threatening asthma exacerbations while on appropriate anti-asthmatic medications.
* Participant has an active bacterial, viral, or helminth parasitic infections; OR a history of ongoing, recurrent severe infections requiring systemic antibiotics
* Participant with a known or suspected underlying immunodeficiency or immune-compromised state as determined by the investigator.
* Participant has a concurrent or recent history of severe, progressive, or uncontrolled renal, hepatic, hematological, intestinal, metabolic, endocrine, pulmonary, cardiovascular, or neurological disease.
* Known active hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or positive HIV serology at the time of screening for subjects determined by the investigators to be at high-risk for this disease.
* Participant has a suspected or active lymphoproliferative disorder or malignancy; OR a history of malignancy within 5 years before the Baseline assessment, except for completely treated in situ non-melanoma skin and cervical cancers without evidence of metastasis.
* Participant has received a live attenuated vaccine ≤ 28 days prior to study randomization.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, oral JAK inhibitor (tofacitinib, ruxolitinib, baricitinib, ritlecitinib, or investigational oral JAK Inhibitors) or ultraviolet (UV) phototherapy with/without Psoralen Ultraviolet A (PUVA) therapy, within 4 weeks prior to the Week 0/Baseline visit
* Participant has been previously treated with dupilumab
* Participant has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus within 1 week before the Baseline visit.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Severity of Alopecia Tool (SALT) score | Baseline and Week 48
  Change in the SALT score from baseline compared to Week 48 in Dupilumab treated vs placebo treated subjects. SALT score is the sum of percentage of hair loss in all areas (higher score indicates greater hair loss). The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time SALT - Scalp divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). Percentage of hair loss in these areas is multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all areas. SALT scores range from 0 (no hair loss) to 100 (complete scalp hair loss) with lower score indicating better health outcomes/less hair loss.

SECONDARY OUTCOMES:
Proportion of participants achieving an absolute SALT score of ≤ 20 at Week 48 in dupilumab vs. placebo-treated participants | Baseline and Week 48
  The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time. The scalp is divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). The percentage of hair loss in these areas is multiplied by the percent surface area of the scalp in that area. The SALT score is the sum of the percentage of hair loss in all areas. The SALT score ranges from 0 (no hair loss) to 100 (complete scalp hair loss), with a lower score indicating better health outcomes/less hair loss.
Change in SALT score in each treatment group at Weeks 48 and 96 compared to baseline | Baseline Week 48 and Week 96
  The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time. The scalp is divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). The percentage of hair loss in these areas is multiplied by the percent surface area of the scalp in that area. The SALT score is the sum of the percentage of hair loss in all areas. The SALT score ranges from 0 (no hair loss) to 100 (complete scalp hair loss), with a lower score indicating better health outcomes/less hair loss.
Proportion of subjects achieving an absolute SALT score of ≤ 20 at Week 48 and Week 96 in each treatment group | Weeks 48 and 96
  The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time. The scalp is divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). The percentage of hair loss in these areas is multiplied by the percent surface area of the scalp in that area. The SALT score is the sum of the percentage of hair loss in all areas. The SALT score ranges from 0 (no hair loss) to 100 (complete scalp hair loss), with a lower score indicating better health outcomes/less hair loss.
Proportion of participants achieving at least 30%/50%/75%/90% improvement (SALT 30/50/75/90) at Week 48 in dupilumab vs. placebo-treated participants | Week 48
  The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time. The scalp is divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). The percentage of hair loss in these areas is multiplied by the percent surface area of the scalp in that area. The SALT score is the sum of the percentage of hair loss in all areas. The SALT score ranges from 0 (no hair loss) to 100 (complete scalp hair loss), with a lower score indicating better health outcomes/less hair loss.
Proportion of participants achieving at least 30%/50%/75%/90% improvement (SALT 30/50/75/90) at Weeks 48 and 96 in each treatment group | Weeks 48 and 96
  The SALT is a validated instrument for measuring the amount of scalp hair loss at a single point in time. The scalp is divided into four areas: vertex (40% of scalp surface area), right profile (18% of scalp surface area), left profile (18% of scalp surface area), and posterior scalp (24% of scalp surface area). The percentage of hair loss in these areas is multiplied by the percent surface area of the scalp in that area. The SALT score is the sum of the percentage of hair loss in all areas. The SALT score ranges from 0 (no hair loss) to 100 (complete scalp hair loss), with a lower score indicating better health outcomes/less hair loss.
Change in Alopecia Areata Symptom Impact Scale (AASIS) from Week 0/Baseline at Week 48 in dupilumab vs. placebo-treated participants | Week 48
  The AASIS is a 13-item, disease specific measure that asks patients with AA about the severity of their symptoms and how these symptoms interfere with their daily functioning. The AASIS uses a 0-10 numeric rating scale that patients find simple to understand and that is easily translated into different languages. AASIS scale 0-10: 0 indicates the symptom was not present and 10 indicates the symptom was as bad as one can imagine, where higher scores indicate worse symptoms.
Change in Alopecia Areata Symptom Impact Scale (AASIS) from Week 0/Baseline at Weeks 48 and 96 in each treatment group | Weeks 48 and 96
  The AASIS is a 13-item, disease specific measure that asks patients with AA about the severity of their symptoms and how these symptoms interfere with their daily functioning. The AASIS uses a 0-10 numeric rating scale that patients find simple to understand and that is easily translated into different languages. AASIS scale 0-10: 0 indicates the symptom was not present and 10 indicates the symptom was as bad as one can imagine, where higher scores indicate worse symptoms.
Patient's Global Impression of Change (PGIC) Scale score at Week 48 in dupilumab vs. placebo-treated subjects | Week 48
  PGIC is a self-administered questionnaire evaluating improvement or worsening of the participant's alopecia areata as compared to the start of the study and uses a single item, "Since the start of the study, my alopecia areata has…", with 7 responses ranging from 0 "no change or worse" to 7 "a great deal better" where higher scores indicate greater improvement.
Patient's Global Impression of Change (PGIC) Scale score at Week 48 and 96 in each treatment group | Weeks 48 and 96
  PGIC is a self-administered questionnaire evaluating improvement or worsening of the participant's alopecia areata as compared to the start of the study and uses a single item, "Since the start of the study, my alopecia areata has…", with 7 responses ranging from 0 "no change or worse" to 7 "a great deal better" where higher scores indicate greater improvement.
Proportion of subjects achieving Alopecia Areata Physician's Global Assessment (aaPGA) = 0-1 at Week 48 in dupilumab vs placebo-treated subjects | Week 48
  The proportion of alopecia areata subjects with aaPGA score of 0 or 1 at Week 48. The aaPGA is used to assess the clinical response to treatment based on a 6-point scale ranging from 0 (no regrowth) to 5 (100% regrowth), where higher scores indicate greater hair regrowth.
Proportion of subjects achieving Alopecia Areata Physician's Global Assessment (aaPGA) = 0-1 at Week 48 and 96 in each treatment group | Weeks 48 and 96
  The proportion of alopecia areata subjects with aaPGA score of 0 or 1 at Week 48. The aaPGA is used to assess the clinical response to treatment based on a 6-point scale ranging from 0 (no regrowth) to 5 (100% regrowth), where higher scores indicate greater hair regrowth.
Number of adverse events reported | Week 96
  Number of adverse events reported throughout the study. The adverse event will be described and categorized as treatment emergent, serious, abnormal in vital signs, and abnormal in lab parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman-Yassky, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - University of California, Irvine, Irvine, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Immediately after publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.